CLINICAL TRIAL: NCT01593319
Title: Is Regional Anesthesia of the Hip Preferable Over Traditional Analgesia in the Acute Stage of the Management of Patients With a Fracture of the Hip
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Landstinget i Värmland (Other)
Responsible Party: Principal Investigator, Panagiotis Tsagkozis, MD, PhD, Landstinget i Värmland
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: NAROP11; 2011-003326-27 (EudraCT Number)
Record Dates: First submitted 2012-04-30; First posted 2012-05-08 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ropivacaine (Active Comparator)
  Interventions: Drug: Ropivacaine
- Natrium chloride (Placebo Comparator)
  Interventions: Drug: Natrium chloride

INTERVENTIONS:
Drug: Ropivacaine — Local injection (fascia iliaca block) using 150 mg ropivacaine
  Other Names: Narop
  Arms: ropivacaine
Drug: Natrium chloride — Placebo injection of Natrium chloride solution
  Arms: Natrium chloride

SUMMARY:
The main hypothesis of the study is that anaesthesia of the hip using infiltration with a local anesthetic solution is preferable over traditional analgesia with oral opioid medications in the acute stage of the management of patients with a fracture of the hip.

To study the hypothesis the investigators designed a prospective randomised study where patients are assigned in two groups, the first receiving local hip anesthesia and the other placebo treatment. Both groups are eligible to use of standard oral pain treatment.

Effect of analgesia as well as medical complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* fracture of the hip

Exclusion Criteria:

* multiple fractures,
* delay (more than 12 hours) from the time of injury until admission to the hospital,
* local infections, hypersensitivity to local analgetics,
* cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Pain | 3 hours

SECONDARY OUTCOMES:
medical complications (Number of participants that develop pressure ulcers, number of participants that develop pneumonia) | under hospitalization (expected average of 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Hallberg, Forskningsschef, Study Chair — Centrum för klinisk forskning. Centralsjukhuset, 651 85 Karlstad, Sweden
Locations (1):
- Ortopedkliniken, Centralsjukhuset i Karlstad, Karlstad, Värmland County, Sweden

REFERENCES:
- [Result] Brisbane Orthopaedic & Sports Medicine Centre Writing Committee; McMeniman TJ, McMeniman PJ, Myers PT, Hayes DA, Cavdarski A, Wong MS, Wilson AJ, Jones MA, Watts MC. Femoral nerve block vs fascia iliaca block for total knee arthroplasty postoperative pain control: a prospective, randomized controlled trial. J Arthroplasty. 2010 Dec;25(8):1246-9. doi: 10.1016/j.arth.2009.11.018. Epub 2010 Feb 23. PMID 20178889
- [Result] Candal-Couto JJ, McVie JL, Haslam N, Innes AR, Rushmer J. Pre-operative analgesia for patients with femoral neck fractures using a modified fascia iliaca block technique. Injury. 2005 Apr;36(4):505-10. doi: 10.1016/j.injury.2004.10.015. PMID 15755432
- [Result] Fletcher AK, Rigby AS, Heyes FL. Three-in-one femoral nerve block as analgesia for fractured neck of femur in the emergency department: a randomized, controlled trial. Ann Emerg Med. 2003 Feb;41(2):227-33. doi: 10.1067/mem.2003.51. PMID 12548273
- [Result] Foss NB, Kristensen BB, Bundgaard M, Bak M, Heiring C, Virkelyst C, Hougaard S, Kehlet H. Fascia iliaca compartment blockade for acute pain control in hip fracture patients: a randomized, placebo-controlled trial. Anesthesiology. 2007 Apr;106(4):773-8. doi: 10.1097/01.anes.0000264764.56544.d2. PMID 17413915
- [Result] Hogh A, Dremstrup L, Jensen SS, Lindholt J. Fascia iliaca compartment block performed by junior registrars as a supplement to pre-operative analgesia for patients with hip fracture. Strategies Trauma Limb Reconstr. 2008 Sep;3(2):65-70. doi: 10.1007/s11751-008-0037-9. Epub 2008 Sep 2. PMID 18762870
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043